CLINICAL TRIAL: NCT02266641
Title: Parental One-carbon Folate and Choline Nutrition Modulates Risk of Off-spring Cancer Development: Human Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201401034RINB
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2017-05

CONDITIONS: Off-spring Cancer Risk
Keywords: one-carbon metabolism; folate; choline; DNA methylation; imprint marker; cancer risks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- healthy pregnant women (Active Comparator): Supply nutrition counseling and multivitamin supplement to people with poor nutritional status
  Interventions: Behavioral: nutrition counseling; Dietary Supplement: multivitamin supplement
- healthy pregnant women's lineal relative with cancer (Experimental): Supply nutrition counseling and multivitamin supplement to people with poor nutritional status
  Interventions: Behavioral: nutrition counseling; Dietary Supplement: multivitamin supplement
- pregnant women or lineal relative with overweight/obesity (Experimental): Supply nutrition counseling and multivitamin supplement to people with poor nutritional status
  Interventions: Behavioral: nutrition counseling; Dietary Supplement: multivitamin supplement
- healthy pregnant women's lineal relative with diabetes (No Intervention): Supply nutrition counseling and multivitamin supplement to people with poor nutritional status

INTERVENTIONS:
Behavioral: nutrition counseling — Pregnancy diet (include one-carbon nutrients)
  Arms: healthy pregnant women; healthy pregnant women's lineal relative with cancer; pregnant women or lineal relative with overweight/obesity
Dietary Supplement: multivitamin supplement
  Arms: healthy pregnant women; healthy pregnant women's lineal relative with cancer; pregnant women or lineal relative with overweight/obesity

SUMMARY:
Parental one-carbon nutrient intake (folic acid and choline) and the genetic polymorphisms of one-carbon metabolic enzyme were interact with regulating embryonic one-carbon metabolic environment, affect fetal DNA and RNA biosynthesis and methyl modification of the genome molecule, to promote the individual nutrient growth factor of growth and development. Inadequate maternal one-carbon nutrient intake combined with genetic polymorphisms of one-carbon enzymatic mutation, causing one-carbon malnutrition, change fetal methyl metabolic nutrition environment. It not only leads to fetal growth mutation - such as folate and choline deficiency, increasing the risk of fetal neural tube defect but also induce abnormal modifying of fetuses's post-genomic methylation markers, may alter imprinted genes function of progenitors, recompile threshold sensitivity or domain in regulation of metabolic reactions of offspring, resulting in long-lasting effect, increasing the risk of chronic diseases of offspring such as cancer. According to the National Nutrition Survey results show that a considerable proportion of the Taiwanese people had poor one-carbon nutritional status. 48% of women intake 66% below the recommended intake reference value of folate. Whether inadequate parental one-carbon nutrients intake combined with genetic polymorphisms of one-carbon enzymatic mutation will cause one-carbon malnutrition of fetus, affecting fetal growth and modifying the risk of cancer development relationship of offspring. It is due to the lack of local ethnic data and empirical scientific reference at home and abroad, so it can not plan an effective maternal and children nutrient education and prevention strategies about methyl nutrition for early cancer prevention for Taiwanese. Therefore, indigenous people is the intended population of study in this project, screening of healthy pregnant women with high risk factor for cancer and obese pregnant women, and detection of one-carbon nutrient intake and biochemical assessment of the nutritional status of the study group. Supplying nutrition education intervention or multivitamin supplement to improve the poor nutritional status of persons. Using related DNA methylation imprint marker about offspring growth and modifying development of cancer as assessment, this project explores the appropriate one-carbon nutrient intake in parents and children and the assessments in regulation of growth and reducing the cancer-related risk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women aged 21-40 years with first and single fetal pregnancy
2. Healthy pregnant women aged 21-40 years with first and single fetal pregnancy and lineal relative had diabetes
3. Healthy pregnant women aged 21-40 years with first and single fetal pregnancy and lineal relative had cancer
4. Healthy pregnant women, who are overweight/obesity (pre-pregnancy BMI≧24 kg/m2) or her lineal relative with overweight/obesity, aged 21-40 years with first and single fetal pregnancy.

Exclusion Criteria:

* Pregnant women who had heart disease, kidney disease, cancer or accepting medical treatment

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Assessment of maternal one-carbon nutrient (folate, choline, betaine, Vitamine B12) intake at the first trimester visit of pregnancy | 7-10 weeks
  Using semiquantitative food frequency questionnaires (FFQ) to calculate dietary intake of one-carbon nutrient
Assessment of maternal one-carbon nutrient (folate, choline, betaine, Vitamine B12) intake at the second trimester of pregnancy | 20-28 weeks
  Using 24 hours dietary recall and dietary record to calculate dietary intake of one-carbon nutrient
Assessment of maternal one-carbon nutrient (folate, choline, betaine, Vitamine B12) intake at the third trimester of pregnancy | 36-37 weeks
  Using 24 hours dietary recall and dietary record to calculate dietary intake of one-carbon nutrient

SECONDARY OUTCOMES:
Measure maternal blood and urine biochemistry (folate, choline, betaine, homocysteine, Vitamine B2, Vitamine B6, Vitamine B12, etc.) | 7-10 weeks
Measure maternal blood imprinted genes (sonic hedgehog, insulin-like growth factor 2, long interspersed nuclear element 1, etc.) DNA methylation status, DNA 8-Hydroxydeoxyguanosine (8-OHdG) and inflammatory markers (TNF-α, NF-κB, Interleukin, etc.) | 7-10 weeks
Measure maternal blood and urine biochemistry (folate, choline, betaine, homocysteine, Vitamine B2, Vitamine B6, Vitamine B12, etc.) | 24-28 weeks
Measure maternal blood imprinted genes (sonic hedgehog, insulin-like growth factor 2, long interspersed nuclear element 1, etc.) DNA methylation status, DNA 8-Hydroxydeoxyguanosine and inflammatory markers (TNF-α, NF-κB, Interleukin, etc.) | 24-28 weeks
Measure maternal blood, cord blood and urine biochemistry (folate, choline, betaine, homocysteine, Vitamine B2, Vitamine B6, Vitamine B12, etc.) | 37-40 weeks
Measure maternal and cord blood and placenta tissues MTHFR C677T genotypes | 37-40 weeks
Measure maternal blood imprinted genes (sonic hedgehog, insulin-like growth factor 2, long interspersed nuclear element 1, etc.) DNA methylation status, DNA 8-Hydroxydeoxyguanosine (8-OHdG) and inflammatory markers (TNF-α, NF-κB, Interleukin, etc.) | 37-40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Nan Lee, Principal Investigator — National Taiwan University Hospital; Kuang-Ta Huang, Principal Investigator — Hueishin women and children clinic; Chin-Pao Cheng, Principal Investigator — National Taiwan University Hospital; Rwei-Fen S. Huang, Principal Investigator — Fu Jen Catholic University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan